CLINICAL TRIAL: NCT00417001
Title: Reduction of Conscious Sedation Requirements by Olfactory Stimulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit participants
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: P05-075
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Colon Cancer Screening; Colon Polyps
Keywords: sedation; colonoscopy; Aroma therapy
MeSH Terms: conditions — Colonic Polyps | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Aroma therapy

SUMMARY:
Colonoscopy for investigation of lower gastrointestinal complaints or for colon cancer screening is one of the more frequent procedures performed by the Divisions of General Surgery and Gastroenterology. Traditionally, this has been performed while under conscious sedation (medication induced) which may improve patient acceptance and tolerance of the procedure but adds to the operative risk of the procedure. The investigators propose a randomized prospective blinded trial to assess the utility of adding pleasing olfactory stimulation to the inhaled oxygen during the conscious sedation for colonoscopy in an effort to reduce the total doses of sedatives required while maintaining a similar level of sedation. This may decrease the overall period of recovery for the patient, increase the number of procedures which may be accomplished, and decrease the potential complications related to conscious sedation.

DETAILED DESCRIPTION:
4. RESEARCH DESIGN/METHODS/SUBJECT JUSTIFICATION

1. General Approach Two hundred and eighty four patients presenting to the endoscopy clinic will be offered participation in the study. They will be randomized to either 1 ml of sterile water or 1 ml of cherry scented flavoring (Lorann Oils Inc, Lansing MI) (identical oil used by our pediatric anesthesiologists for scenting the anesthesia mask during the induction phase of general anesthesia). These will be connected to the inline oxygen tubing via an Leukens trap with oxygen flowing at 4 liters/ minute rate and titrated to maintain a pulse oximetry saturation level of over 90%. The water or flavoring will not be nebulized into the oxygen. The oxygen will pass through the inactive Leukens trap container and pick up whatever aroma is present. A BIS monitor (Aspect Medical Systems Newton MA) will be applied. Data will be recorded at 5 minute intervals (BIS scores). The BIS score will not be used to titrate the sedative medications since the literature is controversial as to whether a given BIS score is consistently considered adequate sedation. Total recovery time (post procedure), BIS scores, and sedative doses will be recorded.

   1. Research Objective To determine if the addition of pleasing olfactory stimulation can reduce the total dose required for sedatives, decrease the recovery time required but maintain the same levels of sedation.
   2. Detail how many groups or arms are in the study and what each receives ' Two groups will be used. One will receive inhalation of cherry flavored essential oil and the other sterile water.
   3. Randomization Procedures A computer generated block randomized schedule will be used. The patients will be randomized the day of the procedure.
2. Methods and Materials Two hundred and eighty four consecutive patients presenting for elective colonoscopy with endoscopist provided sedation (ASA 1 and 2 per NMCP policy) will be offered participation in the trial. They will be consented the day of the procedure by one of the subinvestigators and randomized to either receive olfactory stimulation by cherry flavored oil (via in line aerosol chamber similar to nebulizer treatments) or sterile water. A standard volume of 1 ml will be placed in the chamber without additional water. A BIS monitor will be placed and BIS scores recorded at time zero (prior to sedation) and every 5 minutes during the procedure. The BIS score will not be used to titrate sedation rather the clinical parameters used by the endoscopist will be used (pulse oximetry, blood pressure, heart rate, clinical level of arousal) because it is controversial in the literature using BIS scores to titrate conscious sedation. The BIS scores will provide an additional rough estimate as to the equivalence of levels of sedation during the procedure. Total doses of medications, BIS scores, procedure duration, and recovery duration will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient's presenting for colon cancer screening, colon cancer follow up colonoscopy, or polyp follow up colonoscopy

Exclusion Criteria:

* Allergy to Demerol or Versed, symptomatic colon disease, allergy to a component in the aroma

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2008-01 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Lucha, DO, Principal Investigator — Naval Medical Center Department of Surgery- Portsmouth, VA
Locations (1):
- Naval Medical Center Department of Surgery, Portsmouth, Virginia, United States